CLINICAL TRIAL: NCT02009345
Title: Familial Hypercholesterolemia Canada / Hypercholesterolemie Familiale Canada
Acronym: FHCanada
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Amgen (Industry); Sanofi (Industry); Pfizer (Industry); Merck Sharp & Dohme LLC (Industry); Valeant Canada Limited (Industry); Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Jacques Genest, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: FH Canada
Record Dates: First submitted 2013-11-21; First posted 2013-12-12 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Familial Hypercholesterolemia; Lipid Disorder
Keywords: Familial hypercholesterolemia,; High LDL-cholesterol; Registry; Coronary artery disease
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Lipid Metabolism Disorders; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Plasma and Buffy coat for DNA extraction DNA stock samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Familial hypercholesterolemia (FH) is the most frequent genetic lipoprotein disorder associated with premature CAD. In Canada, the burden of disease is estimated to be approximately 83,500 patients. The goal of this initiative is to create a registry of subjects with FH across Canada. Rare diseases of lipoprotein metabolism are also included. Using a "hub and spoke" model, the registry extends in various communities to link primary care physicians with provincial academic centers. The registry includes clinical, biochemical and demographic information. Specimens (plasma/serum and DNA) are collected for biobanking. The "local" portion of the registry is available for clinicians to manage patient care, and identify relatives for screening and treatment (cascade screening). The Canada-wide registry, which is completely anonymized, will be made available to provide advice to general practitioners and to support collaborative studies in biomedical, clinical, health outcomes and health economics research. The data extracted for the provincial portion of the database will allow administrative database research that will provide important information to key stakeholders and permit allocation of resources. It will also allow a sound and uniform rationale for the use of novel therapeutic agents and provide expert advice to regulatory agencies. At the Canadian level, the database will allow clinicians and researchers to determine the burden of disease and the long-term effects of treatment. Through the creation of a Canada-wide network of academic clinics, integrating lipid specialists, endocrinologists and cardiologists, the Canadian FH registry will lead to significant benefits for FH patients, clinicians and researchers, biopharmaceutical industry and government.

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is a genetic lipoprotein disorder characterized by elevations in low-density lipoprotein cholesterol (LDL-C) >95th percentile for age and gender. Affected individuals may show clinical manifestations (xanthomas, xanthelasmas and premature arcus corneus) although these manifestations are seen less frequently with early diagnosis and treatment. Untreated, FH will lead to atherosclerotic cardiovascular disease (CVD), primarily coronary artery disease (CAD). There are at least three accepted definitions for FH, based on absolute LDL-C levels (MedPed criteria), the Simon-Broome criteria include a fixed cut-point for LDL-C, the presence of DNA mutations and xanthomas and the FH Dutch Criteria (the Netherlands).

There are well-developed FH Registries in the Netherlands, United Kingdom, Spain, France, and the US, through the newly established US FH Foundation. In the United Kingdom, a report on the economic advantages of treating FH revealed that lipid-lowering statin therapy would lead to 101 fewer cardiovascular deaths/1000 patients with FH given treatment. The cost saving from cardiovascular events is estimated at over $CAN 592 million in the UK if all relatives of index cases were identified and treated, compared with no treatment given. This cascade testing strategy has been successfully applied in the Netherlands in families of FH probands with a detected mutation, thus allowing statin treatment of family members at risk of early coronary heart disease.

In Canada, the burden of disease is estimated to be approximately 120,000 patients, based on an allele frequency of LDL-R mutations of 1/311. In the province of Quebec, the allele frequency is approximately 1/270 and the number of affected subjects is approximately 29,000. Left untreated, FH men develop cardiovascular disease (CVD) in the third decade of life and women, in the fourth decade. When identified and treated early, life expectancy is normal.

The purpose of this initiative is to create a registry of subjects with FH across Canada designed to identify subjects with FH and to improve health and healthcare delivery. Rare diseases of lipoprotein metabolism (orphan diseases) are also included (SMASH registry; Systems and Molecular Approach of Severe Hyperlipidemia). This registry includes clinical, biochemical and demographic information. Specimens (plasma/serum and DNA) are collected for biobanking. The "local" portion of the registry is available for clinicians to manage patient care, and identify relatives for screening and treatment (cascade screening). The Canada-wide registry, which is completely anonymized, will be made available to provide advice to general practitioners and to support collaborative studies in biomedical, clinical, health outcomes and health economics research. Access to anonymized data from the registry will be given to researchers, clinicians, biopharmaceutical industry and government by peer-reviewed process.

The Mission of the Canadian FH Registry is to bring together a multi-disciplinary group of physicians, basic and clinical researchers to improve the delivery of care to patients with severe lipoprotein disorders, especially FH, and to foster collaborative research. Our Vision is to create a Canada-wide network of academic clinics, integrating lipid specialists, endocrinologists and cardiologists to treat patients with the highest standard of care and to create a collaborative research environment. Using a "hub and spoke" model, the registry extends in various communities to link primary care physicians with provincial academic centers. The Goals are to improve care to patients with FH and to reduce cardiovascular disease in this population at high risk.

Given the wide geographic distribution of patients with FH, we provide a "hub and spoke" model specialized care. The hubs are based in each province in centers recognized at the national level for their expertise in lipoprotein disorders and with advanced laboratory facilities (medical biochemistry, specialized assays, ultracentrifugation, genetic testing). Radiating from these centers are clinics that treat patients with FH. We propose a three-tier registry (local, provincial and Canada-wide). The local database is nominative, used solely by the clinic or center and contain the information obtained by the local investigators and used for clinical purposes. The provincial database is de-identified and will be used to generate province-specific health outcomes, resource utilization, health economics and comparative epidemiological/genetic/clinical features across provinces. The Canadian database is also anonymous and will serve to generate country-wide statistics, public awareness and research collaborations.

All procedures related to the FH registry are standardized. The various steps associated with the inclusion of patients within the FH Registry are the following: subject with high LDL-C, secondary causes ruled out, FH Criteria satisfied, consent form signed, clinical evaluation, baseline lipid profile, demographic info, family history, longitudinal follow-up (annual data capture). If a patient has a family history of FH, then we start cascade screening. If the FH criteria are not satisfied at the beginning of the study then the patient is being asked to enter in the SMASH registry for other severe disorders of the lipid metabolism. DNA isolation and banking is being performed at individual sites (locally) only. Central biobanking is not possible for now. The question form mainly includes data on the familial history of elevated cholesterol levels and CVD, the patient's medical and surgical history, the physical signs of FH, and the patient's medication profile.

The James Hogg Research Centre at St-Paul's Hospital, UBC, Vancouver is providing the iCAPTURE platform to be used to capture the data from the FH Canada Registry. This center maintains multi-level security for all database and computer systems. The security measures include physical entry to the compute facility and access to the systems within the facility. The server facility is a single entry electronically card accessible room that is equipped with video surveillance. Entry is accessible to the authorized personnel only. All hard drive storage is maintained on a SAN which has data encryption. The database utilizes an Oracle backend and is firewalled and maintained in a separate non public network, and it is FDA (US Food and Drug administration), Health Canada, PHIA (Personal Health Information Act) and PIPEDA (Canada Personal Information Protection and Electronic Documents Act) compliant. All data is de-identified based on role based access and redacted automatically within the database. All user access is logged. A unique identifier is assigned to each patient entered in the database, and parents, siblings and all first-degree relatives of each subject is entered with a distinct identifier. Completely anonymous data, without any identifier -such as hospital ID number, date of birth, family relationships will be made available to researchers, policy makers, governments and industry on a per need basis after a submission of a written request and approval by the Scientific Board in consultation with the Advisory Board.

Potential benefits Patients. Patients will have access to expert care in the field of lipoprotein disorders and CVD prevention. In many cases, optimal treatment of severe hypercholesterolemia may be best provided by experts in the field. They will have access to on-going clinical trials and to novel therapies. Furthermore, individual patients will be offered family screening to identify affected members who would benefit from early diagnosis and treatment. The identification of new FH cases by cascade screening proves to be both cost-effective and aligns with the aim of providing personalized medicine for patients with severe lipoprotein disorders.

Clinicians. The registry will provide the local (i.e. clinic or hospital) framework to diagnose patients according to accepted international criteria for FH, to follow the subjects in time and to perform cascade screening (first, second and third-degree relatives), a cost-effective strategy to screen potentially affected subjects. The registry will also link clinicians into a network of specialized clinics that favor collaborative investigator-initiated research and participation in multi-center studies. The availability of biobanking will allow the storage of plasma/serum and DNA for future research.

Biomedical researchers. The identification of novel genes for FH and other rare lipoprotein disorders has led to a better understanding of metabolic pathways and eventually the potential for novel therapeutic targets. In addition, gene-gene and gene-environment interactions research may shed light on mechanisms of disease. clinical-scientists will have the opportunity to develop investigator-initiated research, using the pan-Canadian registry and biobanking resources as a platform. Researchers in health outcomes and health economics, social, gender and ethnic research will have access to the database in collaboration with provincial administrative databases.

Biopharmaceutical Industry. The biopharmaceutical industry will have access to a group of lipid experts across Canada, with links internationally, a harmonized database for subjects with FH and rare lipoprotein disorders. They will have access to a network of established clinics with a unified database. Access to the registry database will be provided after review of the intended research. This data will be important in determining health economics.

Government. This initiative will allow the development of clinical practice guidelines, to determine resource allocation according to need, the identification of rare (orphan disease) lipoprotein disorders requiring specific techniques, such as extracorporeal LDL filtration for homozygous FH. The initiative will allow the framework to set-up collaborative research under the peer-review system (HSFC, CIHR). Health outcomes and health economic studies will allow resource allocation and quality control. Finally centralized genetic testing would provide molecular diagnostics in a cost-effective manner, when required. This initiative will dovetail with the CIHR C-CHANGE initiative concerning the harmonization of cardiovascular preventive guidelines in Canada. To data, we are the only country with harmonized CVD prevention guidelines.

Knowledge translation and training. Individual academic institutions with a strong biomedical research commitment will offer undergraduate and graduate-level training in the field of lipid and lipoproteins within a country-wide collaborative research environment. Several centers will offer post-doctoral fellowships for clinicians and PhDs in lipoprotein metabolism, health outcomes and health economics research. This training of highly qualified personnel is expected to contribute to the academic and economic engine of the country. A formal training course, aligned with the National Lipid Association, will provide certification on the treatment of lipoprotein disorders. The establishment of clinical practice guidelines for adult and pediatric patients will enable clinicians to hone their clinical practice to the highest standard. By using well established conferences across Canada, the aim will be to integrate novel knowledge into the yearly conference programs across Canada and to disseminate this information to practicing physicians and health care professionals.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnostic criteria for FH, which are:

  * Family and/or personal history of high cholesterol
  * Family and/or personal history of heart disease
  * Abnormal growth on tendons, accumulation of fatty material in the eye
* Family history of FH
* Severe disorder of cholesterol and other lipids in the blood

Exclusion Criteria:

No exclusion criterion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2013-11; Primary Completion 2025-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with FH | From date of start of the study until date of data analysis (expected December 2025) so within the first 10 years of the regisrtry.
  Absolute Number of patients enrolled in the registry, i.e. number of patients with FH diagnosed in Canada (n = xxx) in 10 years of enrolment.

SECONDARY OUTCOMES:
Prevalence rates of FH in Canada | From date of start of the study until date of data analysis (expected December 2025) so within the first 10 years of the regisrtry.
  % of FH patients (Total number of FH patients/Population of canada*100) in 10 years of enrolment.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Genest, MD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- Research Institute of the McGill University Health Centre: Glen site, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Guerin A, Iatan I, Ruel I, Ngufor LF, Genest J. Genetic testing for familial hypercholesterolemia in Quebec, Canada: a single-centre retrospective cohort study. CMAJ Open. 2023 Aug 22;11(4):E754-E764. doi: 10.9778/cmajo.20220108. Print 2023 Jul-Aug. PMID 37607748